CLINICAL TRIAL: NCT02054208
Title: A Double-blind, Single-center, Phase 1/2a Clinical Trial to Evaluate the Safety and Exploratory Efficacy of Intraventricular Administrations of NEUROSTEM® Versus Placebo Via an Ommaya Reservoir in Patients With Alzheimer's Disease
Brief Title: Safety and Exploratory Efficacy Study of NEUROSTEM® Versus Placebo in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-CR-010
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease
Keywords: human umbilical cord blood derived mesenchymal stem cells; stem cells; alzheimer's disease; cognitive ability; mesenchymal stem cells; cord blood
MeSH Terms: conditions — Alzheimer Disease | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Stage 1: 9 subjects (3 subjects for low dose and 6 subjects for high dose) Stage 2: 36 subjects ( 24 subjects for high dose and 12 subjects for placebo) A total of 45 subjects to be enrolled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEUROSTEM (hUCB-MSCs)- low dose (Experimental): human umbilical cord blood derived mesenchymal stem cells Low dose: 1 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  Interventions: Biological: human umbilical cord blood derived mesenchymal stem cells
- NEUROSTEM (hUCB-MSCs) - high dose (Experimental): human umbilical cord blood derived mesenchymal stem cells High dose: 3 x 10^7 cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  Interventions: Biological: human umbilical cord blood derived mesenchymal stem cells
- Placebo (Placebo Comparator): normal saline 2mL, doses separated by 4 weeks for a total of 3 doses
  Interventions: Other: Normal saline 2mL

INTERVENTIONS:
Biological: human umbilical cord blood derived mesenchymal stem cells — Low dose: 1 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  High dose: 3 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  Other Names: NEUROSTEM
  Arms: NEUROSTEM (hUCB-MSCs) - high dose; NEUROSTEM (hUCB-MSCs)- low dose
Other: Normal saline 2mL — Intraventricular administrations of 2mL Normal Saline at 4 week intervals via an Ommaya Reservoir, for a total of 3 administrations
  Arms: Placebo

SUMMARY:
This combined phase 1/2a clinical trial is to investigate the safety, dose limiting toxicity (DLT), and exploratory efficacy of three repeated intraventricular administrations of NEUROSTEM® (human umbilical cord blood-derived mesenchymal stem cells) versus placebo via an Ommaya reservoir at 4 week intervals in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
The study is divided into the 2 stages: dose-escalation in stage 1 and randomized and multiple-dose cohort parallel design in stage 2.The target population for enrollment in this study is patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
1 stage Inclusion Criteria:

1. Korean male or female at 50 -85 years of age
2. Diagnosis of Probable Alzheimer type according to NINCDS-ADRDA criteria at Visit 1 (Screening)
3. Korea Mini-Mental State Examination (KMMSE) score of 18 - 26 at Visit 1 (Screening)
4. Positive for Amyloid on PIB-PET or Florbetaben PET
5. A subject who is informed of the clinical trial and signs a consent form (if unable to sign, a consent from a legally acceptable representative is required)

2 stage Inclusion Criteria:

1. Korean male or female at 50 -85 years of age
2. Diagnosis of Probable Alzheimer type or mild cognitive impairment due to Alzheimer's disease (stage A) according to NIA-AA criteria at Visit 1(Screening)
3. Korea Mini-Mental State Examination (KMMSE) score of over 18 at Visit 1 (Screening)
4. Positive for Amyloid on Florbetaben PET
5. A subject with neurodegeneration (mild atrophy of the brain) as confirmed by MRI
6. A subject who is informed of the clinical trial and signs a consent form (if unable to sign, a consent from a legally acceptable representative is required)

Exclusion Criteria:

1. Concurrent mental disorder (such as schizophrenia, depression, bi-polar diseases or others) aside from dementia
2. Concurrent dementia as a result of other neurodegenerative disorders (due to infectious disease of the central nervous system such as HIV, syphilis), head injury, Creutzfeld-Jacob disease, Pick's disease, Huntington's disease, or Parkinson's disease
3. Diagnosis of severe white matter hyperintensitivity (WMH) according to CREDOS (Clinical REsearch Center for Dementia of South Korea), which is defined as ≥ 25mm of the deep white matter and ≥ 10mm of the periventricular capping/banding in lengths
4. History of stroke within 3 months prior to study enrollment
5. Severe liver disorder (equivalent to double the normal values of ALT and AST) at Visit 1
6. Severe kidney disorder (serum creatinine ≥1.5mg/dL) at Visit 1
7. Pregnant or lactating females
8. Abnormal Laboratory findings at Visit 1

   * Hemoglobin < 9.5 g/dL for male and <9.0 g/dL for female
   * Total WBC Count < 3000/mm3
   * Total Bilirubin >= 3 mg/dL
9. Suspected active lung disease based on chest X-ray at Visit 1
10. Woman of childbearing age who refuses to practice medically acceptable contraceptive method (post menopausal patient with no menstruation for at least 12 months is considered as infertile)
11. History of screening failure for the clinical trial of NEUROSTEM® in the past 6 months
12. Participation in another clinical trial in the past 3 months prior to the beginning (Week 0) of this clinical trial
13. Bleeding disorder (abnormal blood coagulation test result (i.e. platelet count of < 150,000/mm3, PT ≥ 1.5 INR, or aPTT ≥ 1.5 x control anti-coagulant or anti-platelet, without anticoagulant or anti-platelet therapy)
14. Diagnosis of cancer (of any body system, including brain tumor)
15. Substance/alcohol abuse
16. Contraindicated for any of the tests performed during the clinical trial period (for example, MRI, CT, PET)
17. A subject in whom Ommaya reservoir insertion is considered difficult
18. Whom the principal investigator considers inappropriate for participation in the study due to any reasons other than those listed above

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 24 weeks after the first dose
  Number of subjects with adverse event, number of subjects with normal range of vital signs, mixed lymphocyte reaction result, and laboratory examination result

SECONDARY OUTCOMES:
Change from the baseline in ADAS-Cog | 24 weeks after the first dose
  Alzheimer's Disease assessment Scale-Cognitive Subscale
Change from the baseline in S-IADL | 24 weeks after the first dose
  Seoul Instrumental Activities of Daily Living
Change from the baseline in K-MMSE | 24 weeks after the first dose
  Mini Mental State Exmination Korean version
Change from the baseline in CGA-NPI | 24 weeks from the first dose
  Caregiver-administered Neuropsychiatric Inventory
ADAS-Cog Response Rate | 24 weeks after the first dose
  ADAS-cog response is defined as no worsening (no change or improvement on ADAS-cog score) of the ADAS-cog score at 24 weeks after the first administration compared to the baseline
Change in CDR-SOB | 24 weeks after the first dose
  Clinical Dementia Rating-Sum of Box
Change in Florbetaben-PET | 24 weeks after the first dose
  Florbetaben - Pittsburgh Compound B-positron emission tomography
Change in FDG-PET (CMRglc: regional cerebral metabolic rate for glucose) | 24 weeks after the first dose
  fluorodeoxyglucose positron emission tomography
Change in CIBIC-plus | 24 weeks after the first dose
  The Clinician's Interview Based Impression of Change-plus
Change from baseline in MRI (DTI mapping) | 24 weeks after the first dose
  MRI Analysis
Change from the baseline in CSF biomarkers | 24 weeks after the first dose
  biomakrer analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wonil Oh, MD, PhD, Study Director — Medipost Co Ltd.
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee NK, Jang H, Choi Y, Hwangbo S, Lee S, Lee JI, Kim YJ, Chin J, Chang JW, Seo SW, Son HJ, Choi SJ, Na DL, Kim HJ. Mesenchymal Stem Cells With Adjuvant Dexamethasone in Patients With Alzheimer's Disease: A Phase IIa Trial. Dement Neurocogn Disord. 2025 Oct;24(4):272-285. doi: 10.12779/dnd.2025.24.4.272. Epub 2025 Oct 24. PMID 41220869
- [Derived] Choi Y, Shin S, Son HJ, Lee NH, Myeong SH, Lee C, Jang H, Choi SJ, Kim HJ, Na DL. Identification of potential biomarkers related to mesenchymal stem cell response in patients with Alzheimer's disease. Stem Cell Res Ther. 2023 Jul 19;14(1):178. doi: 10.1186/s13287-023-03410-8. PMID 37468918
- [Derived] Kim HJ, Cho KR, Jang H, Lee NK, Jung YH, Kim JP, Lee JI, Chang JW, Park S, Kim ST, Moon SW, Seo SW, Choi SJ, Na DL. Intracerebroventricular injection of human umbilical cord blood mesenchymal stem cells in patients with Alzheimer's disease dementia: a phase I clinical trial. Alzheimers Res Ther. 2021 Sep 14;13(1):154. doi: 10.1186/s13195-021-00897-2. PMID 34521461
- See also: first-in-man study of NEUROSTEM — http://www.clinicaltrials.gov/ct2/show/NCT01297218?term=neurostem&rank=2